CLINICAL TRIAL: NCT04892368
Title: Prospective Single-centre Randomized Controlled Trial to Evaluate Preoperative Home-based Supervised Exercise Program for Prehabilitation of Frail Elderly Patients Undergoing Major Abdominal Surgery, Against Current Home-based Unsupervised Exercise Program.
Brief Title: Efficacy of Preoperative Prehabilitation With a Home-based Supervised Exercise Program Against an Unsupervised Exercise Program for Frail Elderly Patients Undergoing Major Abdominal Surgery
Acronym: HOME-PREPARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-PREPARE-01
Record Dates: First submitted 2021-05-04; First posted 2021-05-19 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Frail Elderly Syndrome; Frailty; Surgery
Keywords: prehabilitation
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home supervised exercise program (Active Comparator): This group receives standard preoperative physiotherapy education as well a home-exercise instructions. They will also receive 3-4 home visits by physiotherapists between recruitment and surgery, to conduct exercises in their homes.
  Interventions: Other: Home-based supervised exercise program
- Home unsupervised exercise program (No Intervention): This group receives standard preoperative physiotherapy education as well a home-exercise instructions.

INTERVENTIONS:
Other: Home-based supervised exercise program — Combination of aerobic and strength training exercises, in addition to home exercise instructions issued during preoperative physiotherapy education.
  Arms: Home supervised exercise program

SUMMARY:
Singapore's population is ageing, and more elderly people are undergoing elective major surgeries. Frail elderly experience greater functional decline and slower recovery in physical function after surgery compared to non-frail elderly. Preoperative prehabilitation aims to enhance both aerobic capacity and physical strength of elderly to attenuate the post-operative decline in physical function. Singapore General Hospital has a bespoke preoperative program - Prehabilitation for Elderly Frail Patients Undergoing Elective Surgeries (PREPARE), where patients receive physiotherapy education and instructions for home-based unsupervised exercise program (uSEP). A hospital-based supervised exercise program had also been established but the take-up rate was low (7.6%) due to barriers such as cost and accessibility. Perioperative supervised exercise training can effect greater gains in functional capacity and muscle strength compared to no supervision. For the elderly with limited transport options to the hospital, home-based supervised programmes may be more convenient compared to hospital-based supervised programmes, but the former is costlier too. Home-interventions may also empower patients with the skills and confidence to maintain their physical fitness at home, which increases their likelihood of exercising after surgery.

The investigators propose a prospective single-center randomized controlled trial to evaluate the efficacy of preoperative prehabilitation with a home-based supervised exercise program (SEP) for frail elderly patients undergoing major abdominal surgery, compared to the mainstay of clinical practice, which is a home-based uSEP.

ELIGIBILITY:
Inclusion Criteria:

* 1. Elective major abdominal surgery
* 2. Lead time >= 14 days to surgery
* 3. Edmonton Frail Scale total score >= 6 points or Functional performance score (Timed up and Go(TUG)) >= 1 point

Exclusion Criteria:

* 1. Inability to provide written informed consent due to cognitive impairment
* 2. Having Comorbid medical conditions interfering with the ability to perform exercise at home or to complete the testing procedures. These include: i. Unstable cardiac conditions ii. Acute illnesses iii. Patients who are completely unable to walk

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2021-04-10 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Change in functional walking capacity from baseline to just before surgery, as measured using the 6-minute walk distance. | From recruitment to 2-days before surgery
  Distance that the patient can walk in 6 min, along a 15-20m hallway, at a pace that the participants will be tired at the end of the distance. This is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.

SECONDARY OUTCOMES:
30-day in-hospital complications | From day of surgery to 30-days afterwards
  Classified using the Clavien Dindo Classification
Hospital length-of-stay | From day of surgery until discharge, or up to 6 months after surgery, whichever occurs first
  Duration that patient stayed in hospital from day of surgery to discharge either to home or step-down care
Health-related quality of life outcomes (HRQoL) as measured using the 12-Item Short Form Survey (SF-12) | Day of recruitment, 2 days before surgery, 4 weeks, 8 weeks and 6 months postoperative
  SF-12 is a 12-item questionnaire that assesses generic health outcomes from the patient's perspective, and covers eight domains: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional & mental health.
Health-related quality of life outcomes (HRQoL) as measured using the EQ-5D-3L | Day of recruitment, 2 days before surgery, 4 weeks, 8 weeks and 6 months postoperative
  The EQ-5D-3L descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, and extreme problems.
Change in 6-minute walking distance | Day of recruitment, 2 days before surgery, 4 weeks and 8 weeks postoperative
  Distance that the patient can walk in 6 min, along a 15-20m hallway, at a pace that the participants will be tired at the end of the distance. This is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Maximal Inspiratory Pressure (MIP) | Day of recruitment, 2 days before surgery, 4 weeks and 8 weeks postoperative
  The maximal inspiratory pressure reflects the strength of inspiratory muscles.
30-second and 1-minute Sit-to-Stands (STS) | Day of recruitment, 2 days before surgery, 4 weeks and 8 weeks postoperative
  The Sit to Stand test reflects lower-extremity strength and endurance.
Handgrip strength (HGS) | Day of recruitment, 2 days before surgery, 4 weeks and 8 weeks postoperative
  The handgrip strength is a measure of muscular strength or the maximum force/tension generated by one's forearm muscles. It reflects upper body strength and overall strength.

CONTACTS AND LOCATIONS:
Locations (1):
- Eileen Yilin Sim, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No